CLINICAL TRIAL: NCT02569723
Title: Pilot Study of a Carbon 14 Oxaliplatin Microdosing Assay to Predict Exposure and Sensitivity to Oxaliplatin-Based Chemotherapy in Advanced Colorectal Cancer
Brief Title: Oxaliplatin Microdosing Assay in Predicting Exposure and Sensitivity to Oxaliplatin-Based Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Kim (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Edward Kim, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 736253; UCDCC#255 (Other: UC Davis); P30CA093373 (NIH); UCDCC#255 (Other: University of California Davis Comprehensive Cancer Center)
Record Dates: First submitted 2015-07-27; First posted 2015-10-07 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Colon Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- carbon C 14 oxaliplatin and oxaliplatin (Experimental): Patients receive carbon C 14 oxaliplatin microdose IV over 120 minutes. Beginning not more than 4 weeks after the initial carbon C 14 oxaliplatin microdose administration, patients receive FOLFOX6 comprised of leucovorin calcium IV, fluorouracil IV over 2 hours (over 46-48 hours via ambulatory infusion pump on days 1 and 2), and oxaliplatin (contain carbon C 14 microdose course I only) IV over 2 hours on day 1.
  Interventions: Drug: Carbon C 14 Oxaliplatin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Carbon C 14 Oxaliplatin — Intravenous infusion
  Other Names: [14C] Oxaliplatin
Drug: Oxaliplatin — Intravenous infusion
  Other Names: Eloxatin

SUMMARY:
This pilot clinical trial studies how well carbon C 14 oxaliplatin microdosing assay works in predicting exposure and sensitivity to oxaliplatin-based chemotherapy in patients with colorectal cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Carbon C 14 is a radioactive form of carbon, exists in nature and in the body at a low level. Microdose carbon C 14 oxaliplatin diagnostic assay may help doctors understand how well patients respond to treatment and develop individualize oxaliplatin dosing in patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of [14C] (carbon C 14) oxaliplatin microdose as a clinical assay to predict oxaliplatin exposure.

SECONDARY OBJECTIVES:

I. To estimate the degree to which a [14C]oxaliplatin microdose predicts the observed pharmacokinetics of standard dose oxaliplatin.

II. To validate that intrapatient variation of exposure to a [14C]oxaliplatin microdose is less than 5%.

III. To detect the levels of oxaliplatin-deoxyribonucleic acid (DNA) adducts induced by oxaliplatin microdosing in peripheral blood mononuclear cells (PBMCs), and correlate the results with patient response and progression free survival on oxaliplatin-based chemotherapy.

IV. To develop preliminary safety data of [14C]oxaliplatin microdosing for future studies.

OUTLINE:

Patients receive carbon C 14 oxaliplatin microdose intravenously (IV) over 120 minutes. Beginning not more than 4 weeks after the initial carbon C 14 oxaliplatin microdose administration, patients receive FOLFOX comprised of leucovorin calcium IV, fluorouracil IV over 2 hours (over 46-48 hours via ambulatory infusion pump on days 1 and 2), and oxaliplatin (contain carbon C 14 microdose course I only) IV over 2 hours on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic colon or rectal adenocarcinoma
* Intent to treat the patient with a leucovorin calcium, fluorouracil, and oxaliplatin (FOLFOX) chemotherapy regimen containing fluorouracil (5-FU), leucovorin, and oxaliplatin according to clinical standard practice; the intent should be to dose oxaliplatin at 85 mg/m^2 on an every 2 week basis
* Treatment with any additional Food and Drug Administration (FDA)-approved biologic agent (i.e. bevacizumab, cetuximab, or panitumumab) is allowed according to standard practice
* Prior radiation or surgery is allowed, but should be finished at least 2 weeks prior to study enrollment; if a participant has prior radiation therapy, at least one measurable lesion outside of the radiation field should be available for the evaluation of response to chemotherapy
* Any number of prior therapies other than oxaliplatin is allowed
* Zubrod performance status equal to or less than 2 (Karnofsky equal to or greater than 50%)
* Life expectancy of at least 3 months
* Absolute neutrophil count greater than or equal to 1,500/microL
* Platelets greater than or equal to 100,000/microL
* Total bilirubin less than 3 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase) less than or equal to 5 x ULN
* Creatinine less than 1.5 x ULN
* Women of child bearing potential must not be pregnant; a pre-study pregnancy test must be negative
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 30 days after study participation
* Men must agree to use adequate contraception (barrier method or abstinence) prior to study entry and for 30 days after study participation
* Ability to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Prior treatment with oxaliplatin
* Patients must not receive concomitant radiation
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Participants who are pregnant or nursing
* Participants who are allergic to any platinum agent
* Participants who have more than grade 1 peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-10-16 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2020-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kim, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carbon C 14 Oxaliplatin and Oxaliplatin
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Carbon C 14 Oxaliplatin and Oxaliplatin
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of 14C Oxaliplatin Microdose as a Clinical Assay to Predict Oxaliplatin Exposure
Description: Correlate area under curve from phase 0 microdosing with area under curve for therapeutic dose of oxaliplatin
Time Frame: 0-5 minutes predose, 5, 15, and 30 minutes, and at 1, 2, 4, 8, and 24 hours after carbon C 14 oxaliplatin microdose
Measure: Number; unit: R squared
Arm/Group | Carbon C 14 Oxaliplatin and Oxaliplatin
Number analyzed (Participants) | 6
R squared | 0.63

2. Secondary Outcome: Duration of Disease Control (DDC) According to RECIST 1.1
Description: Will characterize the repair of DNA adducts in PBMC, using descriptive statistics.
Time Frame: Up to 2 years
Population: Tumor measurements were not collected to assess this outcome measure.
Arm/Group | Carbon C 14 Oxaliplatin and Oxaliplatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events According to CTCAE Version 4
Description: Assess toxicity to both microdoses of carbon C 14 oxaliplatin. Toxicities potentially related to carbon C 14 oxaliplatin will be assessed from initiation of the study to at least 14 days after the administration of the FOLFOX-integrated microdose or until full recover of toxicity (whichever is longer). Safety will be assessed through summaries of adverse events and laboratory evaluations.
Time Frame: Approximately 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carbon C 14 Oxaliplatin and Oxaliplatin
Number analyzed (Participants) | 6
Participants
  Anorexia | 1
  Arthralgia | 1
  Dehydration | 1
  Diarrhea | 2
  Endocrine disorders - Other - Cold sensitivity | 1
  Fatigue | 3
  Hyperkalemia | 1
  Lymphocyte count decreased | 2
  Nausea | 3
  Neutrophil count decreased | 1
  Pain in extremity | 1
  Peripheral sensory neuropathy | 1
  Vomiting | 1
  White blood cell decreased | 1

4. Secondary Outcome: Response Rate Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: Response was determined according to RECIST criteria as either partial response (PR) or one almost complete response (CR) or progressive disease (PD).
Time Frame: Up to 2 years
Population: Tumor measurements were not collected to assess this outcome measure.
Arm/Group | Carbon C 14 Oxaliplatin and Oxaliplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Incidence of Adverse Events According to the Common Terminology Criteria for Adverse Events Version 4
Arm/Group | Carbon C 14 Oxaliplatin and Oxaliplatin
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carbon C 14 Oxaliplatin and Oxaliplatin (N=6)
Anorexia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Endocrine disorders - Other - Cold sensitivity (Endocrine disorders) | 1
Fatigue (General disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Investigations) | 2
Nausea (Gastrointestinal disorders) | 3
Neutrophil count decreased (Investigations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT02569723/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT02569723/ICF_001.pdf